CLINICAL TRIAL: NCT05669222
Title: Functional and Angiography-Derived Strain Guided Multi-Vessel/Lesion Revascularization Strategy in Patients With Acute ST-Segment Elevation Myocardial Infarction (FAVOR V AMI)
Brief Title: The FAVOR V AMI Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FAVOR V AMI
Record Dates: First submitted 2022-12-18; First posted 2022-12-30 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: ST-Segment Elevation Myocardial Infarction; Multivessel Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Quantitative Flow Ratio; ST-Segment Elevation Myocardial Infarction; Multivessel Coronary Artery Disease; Percutaneous Coronary Intervention; Radial Wall Strain
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Angiography; Coronary Angiography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a blinded clinical trial. Subjects and clinical assessor (including the follow-up research personnel, clinical events committee (CEC) members, and angiographic core laboratory analysts) will be blinded to the assignment results. All the study site personnel will receive training for the blinding measures before the trial initiating. In addition to standard procedural sedation, music-playing headphones will be worn by the patient during the whole procedure, and patients in both groups will be preset a 10-minute delay for μQFR+RWS or sham calculation before the PCI procedure, a lesion/device evaluation form is required to fill in during the period in both groups, to reduce the possibility of unblinding. All the study site personnel will be trained not to disclose the treatment assignment to the subject in any unplanned time. Blinding to the subjects will maintain until 5-year follow-up completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST Guided Strategy (μQFR+RWS) (Experimental): 1. μQFR is measured in all non-infarct related arteries containing any non-culprit lesion with visually-assessed DS% ≥50% and ≤90% with RVD ≥2.5 mm.
     1. μQFR ≤0.80: PCI
     2. RWS ≥13%: PCI
     3. μQFR >0.80 and RWS <13%: Deferral
     4. DS% >90%: PCI without the need of μQFR or RWS
  2. For all patients undergoing PCI, post-PCI μQFR measurement is recommended; if μQFR <0.90, if the reason is obvious post-dilation with a non-compliant balloon or bail-out stenting should be considered; if the reason is not obvious intravascular imaging should be considered.
  Interventions: Diagnostic Test: FAST Technique; Diagnostic Test: Angiography
- Standard Treatment Strategy (Sham Comparator): 1. PCI should be performed of all non-culprit lesions with visual DS% ≥70% in all non-infarct related arteries with RVD ≥2.5 mm;
  2. For a non-culprit lesion with visually DS% 50-70%, PCI can be performed if FFR ≤0.80 or iFR ≤0.89.
  Interventions: Diagnostic Test: Angiography

INTERVENTIONS:
Diagnostic Test: FAST Technique — The next-generation QFR (μQFR) introduces a more intelligent algorithm and supports single-projection rapid calculation with a diagnostic accuracy of 93.0% compared with FFR; Computational RWS technique facilitates the assessment of lesion vulnerability.
  Other Names: The next-generation quantitative flow ratio and radial wall strain
  Arms: FAST Guided Strategy (μQFR+RWS)
Diagnostic Test: Angiography — Coronary angiography is a procedure that uses contrast under x-ray pictures to detect stenosis in the coronary arteries.
  Other Names: Coronary angiography

SUMMARY:
The FAVOR V AMI study is a prospective, multicenter, blinded, randomized, sham-controlled trial comparing the long-term clinical outcomes of the "Functional and Angiography-derived Strain inTegration (FAST)" technique (next-generation quantitative flow ratio [μQFR] and radial wall strain [RWS]) guided percutaneous coronary intervention (PCI) strategy, with standard treatment strategy, in patients with ST-segment elevation myocardial infarction (STEMI) and multivessel coronary disease (MVD).

DETAILED DESCRIPTION:
The FAVOR V AMI study is a prospective, multicenter, blinded, randomized, sham-controlled trial comparing the long-term clinical outcome of the two PCI strategies, the FAST guided strategy (test group) versus standard treatment strategy (control group), in a high-risk population with STEMI and MVD who underwent successful primary PCI of the infarct-related artery. The primary endpoint is major adverse cardiac events (MACE), defined as a composite of all-cause death, myocardial infarction (MI), or ischemia-driven revascularization when the last patient reaches 6-month follow-up. The major secondary endpoint is cardiovascular death and MI when at least 395 total events have accrued. The study hypothesis is the FAST (μQFR+RWS) guided PCI strategy is superior to a standard treatment strategy by the primary and major secondary endpoint.

For the patients randomized to μQFR+RWS group, μQFR will be measured in all non-infarct related arteries containing any non-culprit lesion with visually-assessed percentage diameter stenosis (DS%) ≥50% and ≤90% with reference vessel diameter (RVD) ≥2.5 mm. If μQFR ≤0.80 or RWS ≥13%, PCI will be performed; if μQFR >0.80 and RWS <13%, the procedure will deferral; if DS% >90%, PCI should be performed without the need of μQFR or RWS. For all patients undergoing PCI, post-PCI μQFR measurement is recommended; if μQFR <0.90, if the reason is obvious post-dilation with a non-compliant balloon or bail-out stenting should be considered; if the reason is not obvious intravascular imaging should be considered. For the patients randomized to standard treatment group, PCI should be performed of all non-culprit lesions with visual DS% ≥70% in all non-infarct related arteries with RVD ≥2.5 mm; for a non-culprit lesion with visually DS% 50-70%, PCI can be performed if fractional flow reserve (FFR) ≤0.80 or instantaneous wave-free ratio (iFR) ≤0.89. All patients will be followed by either telephone or clinic visit at 1 month, 6 months,1 year, 2 years, 3 years, 4 years and 5 years.

The sample size will be about 5,000 using an event-driven sample calculation. An adaptive design will be implemented for sample size re-estimation when 90% of patients have been enrolled. All principal analyses will take place in the intention-to-treat (ITT) population. The primary and major secondary endpoints will be analyzed in prespecified subgroups, including age (≥65 vs. <65), sex (men vs. women), diabetes (yes vs. no), time from symptom onset to primary PCI (≤ vs. > median), planned number of NCLs for PCI in the control arm (0/1 vs. 2 vs. 3), infarct related artery (LM/LAD vs, others), untreated CTOs with RVD ≥2.5 mm in non-infarct related artery (yes vs. no), timing of elective PCI (same hospitalization as the emergency PCI vs. during an elective readmission), P2Y12 inhibitor therapy (Clopidogrel vs. Ticagrelor), treatment of any non-infarct lesion with DS >90% prior to randomization (yes vs. no), LVEF (echo post primary PCI, prior to randomization) (>40% vs. ≤40%), Killip Class (I vs. ≥II), lesion location of non-culprit lesion (LM/LAD vs. others), diseased vessels (two-vessel disease vs. LM/three-vessel disease), moderate or severe calcification in any NCL (yes vs. no), bifurcation lesion with planned main vessel and SB treatment in any NCL (yes vs. no), intravascular guidance during the randomized procedure (yes vs. no), μQFR grayzone (μQFR < 0.75 vs. = 0.75-0.85 vs. > 0.85 [by core laboratory]), μQFR-based functional SYNTAX score (FSSQFR, low tertile vs. mid tertile vs. high tertile [by core laboratory]), post-PCI μQFR (≥0.90 vs. <0.90 [by core laboratory]), angiography-derived IMR (≥2.5 mmHgs/cm vs. <2.5 mmHgs/cm [by core laboratory]), residual physiology pattern (PPG diffuse vs. local [by core laboratory]), μQFR-based residual functional SYNTAX score (rFSSQFR, 0 vs. ≥ 1 [by core laboratory]), learning experience of μQFR/RWS (first half vs. second half of enrolled cases in each center).

ELIGIBILITY:
Inclusion Criteria:

* General inclusion

  1. Age ≥18 years
  2. STEMI ≤30d
  3. Successful primary PCI of all culprit lesion(s) responsible for the STEMI (visually-assessed residual stenosis <30% in stent-treated lesions or <50% in DCB-treated or PTCA-treated lesions, with TIMI-3 flow in all treated vessels)
  4. No MACE event between the index PCI and the staged randomized procedure
  5. Able to understand the trial design and provide written informed consent
* Angiographic inclusion:

  1. The presence of at least 1 non-culprit lesion with DS% 50%-90% in any non-infarct related artery with RVD ≥2.5 mm by visual assessment
  2. Non-culprit lesions are potentially eligible for PCI Note: All lesions in the infarct related arteries with DS ≥70% and RVD ≥2.5 mm by visual assessment must be successfully treated either during the index primary PCI or the staged procedure prior to randomization Note: There may also be 1 or more NCL with DS% >90% (including a CTO) as long as there is at least 1 NCL with DS% 50%-90% as above. Any such lesions in which PCI is intended must be treated successfully either during the index primary PCI or the staged procedure prior to randomization.

Exclusion Criteria:

* General exclusion

  1. Cardiogenic shock or refractory hypotension (Killip IV)
  2. On pressors or use of or need for intra-aortic balloon pump or other mechanical circulatory support devices
  3. Intubated
  4. Prior thrombolytic therapy for this admission
  5. Cockcroft-Gault-calculated CrCl <30 ml/kg
  6. Pregnant or woman of child-bearing potential
  7. Life expectancy less than 1 year for non-cardiac causes
  8. Allergy to iodine-containing contrast agents which cannot be adequately premedicated
  9. Unable to tolerate DAPT for at least 6 months
  10. Prior CABG or planned CABG
  11. Any planned surgery within 6 months
  12. Any condition that may interfere with any follow-up procedures (e.g. dementia, drug use)
* Angiographic exclusion

  1. Poor angiographic image quality precluding vessel contour detection or with suboptimal contrast opacification, branch ostium cannot be shown clearly, severe overlap in the stenosed segment or severe tortuosity of any interrogated vessel deemed not amenable to μQFR or RWS measurement
  2. Unable to judge culprit lesion or infarct-related artery according to current evidence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events (MACE) | From the date of first randomization until a total number of 395 events of MACE is reached (median follow-up of approximately 1.5 years)
  Defined as a composite of all-cause death, myocardial infarction (MI), or ischemia-driven revascularization

SECONDARY OUTCOMES:
Incidence of cardiovascular death and MI (Major secondary endpoint） | From the date of first randomization until a total number of 395 events of cardiovascular death and MI is reached (median follow-up of approximately 3 years)
  Defined as a composite of cardiovascular death and MI
Rate of lesion success | Immediately post the PCI procedure
  Defined as: 1) angiographic success (core laboratory-assessed residual stenosis <30% in stent-treated lesions or <50% in DCB-treated or PTCA-treated lesions, with TIMI-3 flow in the treated vessel); and 2) physiological success (post-PCI μQFR ≥0.80 assessed by core lab)
Rate of procedural success | Maximum of 7 days
  Defined as lesion success in all treated lesions without in-hospital MACE
Incidence of death | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Including cardiovascular, non-cardiovascular or undetermined
Incidence of all MI | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Including periprocedural MI (SCAI definition) and spontaneous MI (target vessel-related or non-target vessel-related, culprit lesion-related or non-culprit lesion-related)
Incidence of any revascularization | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Including ischemia-driven or non-ischemia driven, target vessel-related or non-target vessel-related, culprit lesion-related or non-culprit lesion-related
Incidence of definite/probable stent thrombosis (ARC-2) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  By ARC-2 definition and including acute, subacute, late and very late stent thrombosis
Angina status evaluation | 6 months, 1 year, 3 years, 5 years
  As assessed by the Seattle Angina Questionnaire (SAQ)
Health-related quality of life evaluation | 6 months, 1 year, 3 years, 5 years
  As assessed by the European Quality of Life-5 Dimensions (EQ-5D)
Cost-effectiveness evaluation | 6 months, 1 year, 3 years, 5 years
  As assessed by the Incremental cost effectiveness ratio (ICER) using the composite endpoint (including myocardial infarction, any revascularization, stent thrombosis, cerebrovascular and major bleeding events)
Cost-utility evaluation | 6 months, 1 year, 3 years, 5 years
  As assessed by the Incremental cost-utility ratio (ICUR) using quality-adjusted life years (QALYs)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Xu, MBBS, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing; Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen; Lei Song, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313
- [Background] Erlinge D, Maehara A, Ben-Yehuda O, Botker HE, Maeng M, Kjoller-Hansen L, Engstrom T, Matsumura M, Crowley A, Dressler O, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Okkels Jensen L, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Muller JE, Stone GW; PROSPECT II Investigators. Identification of vulnerable plaques and patients by intracoronary near-infrared spectroscopy and ultrasound (PROSPECT II): a prospective natural history study. Lancet. 2021 Mar 13;397(10278):985-995. doi: 10.1016/S0140-6736(21)00249-X. PMID 33714389
- [Background] Mehta SR, Wood DA, Storey RF, Mehran R, Bainey KR, Nguyen H, Meeks B, Di Pasquale G, Lopez-Sendon J, Faxon DP, Mauri L, Rao SV, Feldman L, Steg PG, Avezum A, Sheth T, Pinilla-Echeverri N, Moreno R, Campo G, Wrigley B, Kedev S, Sutton A, Oliver R, Rodes-Cabau J, Stankovic G, Welsh R, Lavi S, Cantor WJ, Wang J, Nakamya J, Bangdiwala SI, Cairns JA; COMPLETE Trial Steering Committee and Investigators. Complete Revascularization with Multivessel PCI for Myocardial Infarction. N Engl J Med. 2019 Oct 10;381(15):1411-1421. doi: 10.1056/NEJMoa1907775. Epub 2019 Sep 1. PMID 31475795
- [Background] Puymirat E, Cayla G, Simon T, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, Gallet R, Khalife K, Morelle JF, Motreff P, Lemesle G, Dillinger JG, Lhermusier T, Silvain J, Roule V, Labeque JN, Range G, Ducrocq G, Cottin Y, Blanchard D, Charles Nelson A, De Bruyne B, Chatellier G, Danchin N; FLOWER-MI Study Investigators. Multivessel PCI Guided by FFR or Angiography for Myocardial Infarction. N Engl J Med. 2021 Jul 22;385(4):297-308. doi: 10.1056/NEJMoa2104650. Epub 2021 May 16. PMID 33999545
- [Background] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Background] Tu S, Ding D, Chang Y, Li C, Wijns W, Xu B. Diagnostic accuracy of quantitative flow ratio for assessment of coronary stenosis significance from a single angiographic view: A novel method based on bifurcation fractal law. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:1040-1047. doi: 10.1002/ccd.29592. Epub 2021 Mar 4. PMID 33660921
- [Background] Hong H, Li C, Gutierrez-Chico JL, Wang Z, Huang J, Chu M, Kubo T, Chen L, Wijns W, Tu S. Radial wall strain: a novel angiographic measure of plaque composition and vulnerability. EuroIntervention. 2022 Sep 8;18(12):1001-10. doi: 10.4244/EIJ-D-22-00537. Online ahead of print. PMID 36073027